CLINICAL TRIAL: NCT02289144
Title: Ceritinib in Mutation and Oncogene Directed Therapy in Metastatic or Locally Advanced Anaplastic/Undifferentiated Thyroid Cancer
Brief Title: Ceritinib in Mutation and Oncogene Directed Therapy in Thyroid Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: study was on hold for protocol redesign; decided to not move forward with study.
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 082014-029
Record Dates: First submitted 2014-10-06; First posted 2014-11-13 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-01

CONDITIONS: Metastatic Anaplastic Thyroid Cancer; Locally Advanced Anaplastic, Undifferentiated Thyroid Cancer
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic | interventions — ceritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ceritinib (Experimental)
  Interventions: Drug: Ceritinib

INTERVENTIONS:
Drug: Ceritinib — 750 mg orally daily on day 1. Continue every 4 weeks and every 2 cycles (1 Cycle is 28 days long) : until progression, new recurrence or distant metastasis, as well as enlargment of an existing metastasis on radiological Imaging.

SUMMARY:
This is an, open-label, protocol designed to evaluate the activity of targeted therapy in anaplastic/undifferentiated thyroid cancer. Arm A will evaluate ATC/UTC with mutations or rearrangements detected in the ALK gene.

There is no effective treatment for anaplastic thyroid cancer in the locally recurrent or metastatic setting. Ceritinib will be administered to the patient until disease progression by RECIST 1.1, unacceptable toxicity, withdrawal of consent, or discontinuation of the trial for any other reason.

The primary focus of this arm of the protocol is identifying ceritinib's activity in anaplastic or undifferentiated thyroid cancer patients. Those patients with mutations identified in their ALK gene by sequencing their tumor samples, or with the established ALK abnormalities will be treated with ALK-inhibitors. These include the Ventana assay and Vysis FISH probe, and patients with tumors positive by this assay will also be considered eligible for therapy on the trial.

Therapeutic Portion:

ARM A: ALK Abnormality IND Ceritinib 750 mg orally daily on Day 1 Continue q4 weeks x 2 cycles

Primary Endpoint: The development of progression; new recurrence or distant metastasis, as well as enlargement of an existing metastasis on radiographic imaging.

Secondary Endpoints:

1. Overall response rate for patients treated with ceritinib as part of the study.
2. Death of study participant due to any cause.

DETAILED DESCRIPTION:
This is an, open-label, protocol designed to evaluate the activity of targeted therapy in anaplastic/undifferentiated thyroid cancer. Arm A will evaluate ATC/UTC with mutations or rearrangements detected in the ALK gene.

There is no effective treatment for anaplastic thyroid cancer in the locally recurrent or metastatic setting. Ceritinib will be administered to the patient until disease progression by RECIST 1.1, unacceptable toxicity, withdrawal of consent, or discontinuation of the trial for any other reason.

The primary focus of this arm of the protocol is identifying ceritinib's activity in anaplastic or undifferentiated thyroid cancer patients. Those patients with mutations identified in their ALK gene by sequencing their tumor samples, or with the established ALK abnormalities will be treated with ALK-inhibitors. These include the Ventana assay and Vysis FISH probe, and patients with tumors positive by this assay will also be considered eligible for therapy on the trial.

The goal of this multi-center, multi-arm trial is to measure the impact of treating metastatic anaplastic thyroid cancer patients with targeted therapy selected for these patients due the presence of a genetic mutation or other aberration. This trial will serve as a framework by which new biomarker-drug combinations can be identified and added as new arms.

Therapeutic Portion:

ARM A: ALK Abnormality IND Ceritinib 750 mg orally daily on Day 1 Continue q4 weeks x 2 cycles

Primary Endpoint: The development of progression; new recurrence or distant metastasis, as well as enlargement of an existing metastasis on radiographic imaging. CT scans of the neck, chest, abdomen and pelvis will be performed at baseline and every two cycles (cycles are 28 days long) according to standard of care. Other imaging of these areas such as PET/MRI will be allowed if CT cannot be performed. MRI of the brain will be performed at baseline and as clinically indicated. Wherever it can be safely given, radiographic contrast agents should be given for the imaging studies.

Secondary Endpoints:

1. Overall response rate for patients treated with ceritinib as part of the study.
2. Death of study participant due to any cause.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of anaplastic thyroid cancer or undifferentiated thyroid cancer that demonstrates mutation in the ALK gene as assessed by sequencing of the tumor specimen for Arm A. Other ALK abnormalities as detected by the approved FISH test (Abbott Molecular Inc), using Vysis breakapart probes (defined as 15% or more positive tumor cells); or the Ventana IHC test will also be seen as evidence of ALK abnormality and meeting eligibility requirement.
2. Patients will not have any other curative therapeutic option, such as radiation or surgery.
3. WHO performance status 0-2.
4. Age greater then or equal to 18 years.
5. Patients must have recovered from all toxicities related to prior anticancer therapies to ≤ Grade 2 (CTCAE v 4.03), provided that any concomitant medication is given prior to initiation of treatment with ceritinib. Exception to this criterion: patients with any grade of alopecia are allowed to enter the treatment.
6. Adequate organ function: the following laboratory criteria have been met:

   * Absolute neutrophil count (ANC) greater then or equal to 1.5 x 109/L
   * Hemoglobin (Hgb) ≥ 8 g/dL
   * Platelets greater then or equal to 75 x 109/L
   * Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN), except for patients with Gilbert's syndrome who may be included if total bilirubin ≤ 3.0 x ULN and direct bilirubin ≤ 1.5 x ULN
   * Aspartate transaminase (AST) < 2.0 x ULN, except for patients with liver metastasis, who are only included if AST < 3 x ULN; alanine transaminase (ALT) < 2.0 x ULN, except for patients with liver metastasis, who are only included if ALT < 3 x ULN
   * Calculated or measured creatinine clearance (CrCL) less then or equal to 30 mL/min
7. Patient must have the following laboratory values or have the following laboratory values corrected with supplements to be within normal limits at screening:

   * Potassium ≥ LLN
   * Magnesium ≥ LLN
   * Phosphorus ≥ LLN
   * Total calcium (corrected for serum albumin) ≥ LLN
8. Written informed consent for the protocol must be obtained prior to any screening procedures.
9. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other procedures.

Exclusion Criteria:

* Patients eligible must not meet any of the following criteria:

  1. Patients with known hypersensitivity to any of the excipients of ceritinib (microcrystalline cellulose, mannitol, crospovidone, colloidal silicon dioxide and magnesium stearate).
  2. Patients with symptomatic CNS metastases who are neurologically unstable or have required increasing doses of steroids within the 1 week prior to study entry to manage CNS symptoms.
  3. Prior therapy with ceritinib.
  4. Presence or history of a malignant disease other than thyroid cancer that has been diagnosed and/or required therapy within the past year and is undergoing active anticancer treatment. Exceptions to this exclusion include the following: completely resected basal cell and squamous cell skin cancers, and completely resected carcinoma in situ of any type.
  5. Patients with known history of extensive disseminated bilateral interstitial fibrosis or interstitial lung disease, including a history of pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, obliterative bronchiolitis, and clinically significant radiation pneumonitis (i.e. affecting activities of daily living or requiring therapeutic intervention).
  6. Patient has clinically significant, uncontrolled heart disease and/or recent cardiac event (within 6 months), such as:

     * unstable angina within 6 months prior to screening;
     * myocardial infarction within 6 months prior to screening;
     * history of documented congestive heart failure (New York Heart Association functional classification III-IV);
     * uncontrolled hypertension defined by a Systolic Blood Pressure (SBP) ≥ 160 mm Hg and/or Diastolic Blood Pressure (DBP) ≥ 100 mm Hg, with or without antihypertensive medication
     * initiation or adjustment of antihypertensive medication(s) is allowed prior to screening;
     * ventricular arrhythmias; supraventricular and nodal arrhythmias not controlled with medication;
     * other cardiac arrhythmia not controlled with medication;
     * corrected QTc > 450 msec using Fridericia correction on the screening ECG
  7. Impaired GI function or GI disease that may alter absorption of ceritinib or inability to swallow up to five ceritinib capsules daily.
  8. Ongoing GI adverse events > grade 2 (e.g. nausea, vomiting, or diarrhea) at the start of the study.
  9. Receiving medications that meet one of the following criteria and that cannot be discontinued at least 1 week prior to the start of treatment with ceritinib and for the duration of participation (see Appendix 1 Tables):

     * Medication with a known risk of prolonging the QT interval or inducing Torsades de Pointes (please refer to http://www.azcert.org/medical-pros/drug-lists/drug-lists.cfm)
     * Strong inhibitors or strong inducers of CYP3A4/5 (please refer to http://medicine.iupui.edu/flockhart/table.htm or http://www.druginteractioninfo.org)
     * Medications with a low therapeutic index that are primarily metabolized by CYP3A4/5, CYP2C8 and/or CYP2C9 (please refer to http://medicine.iupui.edu/flockhart/table.htm or http://www.druginteractioninfo.org)
     * Therapeutic doses of warfarin sodium (Coumadin) or any other coumadin-derived anti-coagulant. Anticoagulants not derived from warfarin are allowed (eg, dabigatran, rivaroxaban, apixaban).
     * Unstable or increasing doses of corticosteroids
     * enzyme-inducing anticonvulsive agents
     * herbal supplements
  10. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
  11. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and agree to continue for 3 months after the last dose of study treatment. Highly effective contraception methods include:

      * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
      * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
      * Male sterilization (at least 6 months prior to screening) with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate. For female subjects on the study the vasectomized male partner should be the sole partner for that subject.
      * Combination of any two of the following (a+b or a+c or b+c):

        1. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception.
        2. Placement of an intrauterine device (IUD) or intrauterine system (IUS).
        3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.

      In case of use of oral contraception, women should have been stable on the same pill for a minimum of 3 months before taking study treatment.

      Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to screening. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
  12. Sexually active males unless they agree to use a condom during intercourse while taking drug and agree to continue for 3 months after the last dose of study treatment. Male patients for 3 months should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Development of Progression | Radiographic Imaging Assessments at Screening and every 56 days until evidence of progression (average 7 months) or unacceptable toxicity, withdrawal of Consent, or discontinuation of the trial for any other reason.
  Ceritinib will be administered to the patient until disease progression by RECIST (Response Evaluation Criteria In Solid Tumors).

CONTACTS AND LOCATIONS:
Overall Officials: Saad A Khan, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No